CLINICAL TRIAL: NCT02336295
Title: Developing and Validating a Food Frequency Questionnaires (FFQ) for the Vegan Population in Israel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 0469-14-TLV
Record Dates: First submitted 2015-01-01; First posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Vegan Diet

ARMS (1):
- Food Frequency Questionnaires (Other): Filling out a Food Frequency Questionnaires (FFQ)
  Interventions: Other: Food Frequency Questionnaires

INTERVENTIONS:
Other: Food Frequency Questionnaires — filling a Food Frequency Questionnaires

SUMMARY:
The study aims to validate a Food Frequency Questionnaire (FFQ) designed specifically for the vegan population in Israel. The participants will complete the FFQ, and the data will be verified by evaluating the participants energy expenditure (by measuring BMR, body composition and daily activity) and conducting a 24-hour food interview.

ELIGIBILITY:
Inclusion Criteria:

* consumption of beef, chicken, fish, eggs, milk or dairy is no more than once a month, for the last 6 months
* age 18-40

Exclusion Criteria:

* consumption of beef, chicken, fish, eggs, milk or dairy more than once a month
* chronic conditions (such as diabetes, hypertension, cardiovascular disease)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Daily energy consumption (Kcal/Day) | 24 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Unit, Sourasky Medical Center, Tel Aviv, Israel